NCT : 1690/KEPK/XII/2019

: The Effect of Combination Therapy Using Li-ESWT and PDE-5 Inhibitor Compared to PDE-5 Inhibitor Alone in Patients With Erectile Dysfunction Title

Date : December 1, 2019



